CLINICAL TRIAL: NCT05458570
Title: Ethnic Predisposition, Risk Factors & Breast Cancer Presentation; a 10 Year Data. Single Centered Prospective Cohort Study From Karachi
Brief Title: Ethnic Predisposition, Risk Factors & Breast Cancer Presentation.
Acronym: BC
Status: Completed | Type: Observational
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Mehwish Mooghal , MBBS, Dr Mehwish Mooghal, Bahria University
Other Study IDs: BahriaUni
Record Dates: First submitted 2022-07-09; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer
Keywords: breast cancer susceptibility; breast cancer, familial; breast cancer, right sided; family history; brca1 brca2; ethnicity
MeSH Terms: conditions — Breast Neoplasms; Breast Cancer, Familial; Unilateral Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer: Breast cancer patients presenting to single center in Karachi over the period of 10 years. The aim was to look for ethnic predisposition of population, age of breast cancer, stage at arrival and menopausal status specific to our population. No intervention done.
  Interventions: Other: Breast Cancer positive patients

INTERVENTIONS:
Other: Breast Cancer positive patients

SUMMARY:
Breast cancer, a leading cause of mortality among females, has been the center of research for many decades. Work is in progress to further advance the research worldwide and in our region. This study is conducted to look into regional ethical predilection, clinical presentation/stage, pathological subtypes & risk factors of BC among patients of Karachi, with the aim of proposing a ground to policy making regarding protocol setting for screening and management of BC for our region.

DETAILED DESCRIPTION:
Background Breast cancer, a leading cause of mortality among females, has been the center of research for many decades. Work is in progress to further advance the research worldwide and in our region. This study is conducted to look into regional ethical predilection, clinical presentation/stage, pathological subtypes & risk factors of BC among patients of Karachi, with the aim of proposing a ground to policy making regarding protocol setting for screening and management of BC for our region.

Methods A prospective cohort single-centered study conducted, which included 500 female patients who attended one surgical unit of a tertiary care public hospital Karachi, during the period of 2010 - 2020. The study was performed in line with the principles of the Declaration of Helsinki and data collection started after taking hospital ethical review board's approval because personal data of patients was used. Afterwards, informed written consent was taken from every included patient. Prior to collecting data, all researchers were thoroughly trained with regards to data collection and examination of patients to eliminate observer bias. Non probability consecutive sampling technique was used. The allotted patients were followed by same researcher from presentation till the end of follow up to avoid observer bias; through direct patient interaction in OPDs and wards, radiological and histo-pathological results from investigations performed and regular follow up of patients during the complete disease period. The retrieved information was filled on pre designed pro-forma. Patients were preemptively explained about our reason for collecting data and its implications. The study is reported according to STROCSS 2021 guidelines.15 Our inclusion criteria was ; female sex, age ≥ 20 years, patients with availability of complete clinical details, biopsy proven breast cancer, no previous history of breast cancer treatment from other centers, all regional ethnicities(residents of Karachi, Sindh only) and all stages of breast cancer. Exclusion criteria of the study was; previously treated breast cancer patients, recurrent BC, female ≤19 years, male/transgender, females coming for treatment from other provinces/foreigners.

Thorough history of all patients obtained including relevant risk factors; i-e age, family history of BC, marital status, age at first born baby, parity, age of menarche/menopause, socio-economic status and ethnicity. Detailed physical examination including clinical presentation of breast lump, its size, side (right/left breast) and site, nipple discharge, nipple retraction, skin involvement, fixity to underlying structures, and lymph node status, was carried out in each patient by a single examiner. Patients presenting with a discrete lump, nipple discharge, nipple changes, skin changes, palpable axillary lymph nodes were subjected to further investigation. Ultrasonography and mammogram of the breast, where possible, were performed as initial imaging modality. FNAC/Biopsy, was carried out in all patients to confirm the diagnosis of BC, its subtype and receptors status. For staging; x-ray chest, ultrasound abdomen for liver and pelvis/ CT chest & abdomen were done on case based need. Bone scan was performed in only symptomatic cases. After thorough overall assessment, clinical stage of BC was assigned to each patient, and stage based treatment was carried out in every patient. Patients having localized disease (≤stage 2A) underwent surgical intervention first followed by chemo/radiotherapy, regional disease(≥ stage 2B) had neo-adjuvant followed by surgery, and advanced disease(stage 4) were given palliation.16 Post operatively detailed histological report of specimen and microscopic involvement of the lymph nodes status were also noted.

Primary outcomes of the cohort were age, ethnicity, family history, stage/histological type and menopausal status while secondary outcomes were parity, marriage, symptoms, lump size/site and socioeconomic status. After collecting the required data on pro forma, it was analyzed using descriptive statistics by SPSS version 23.0 software. With sample size of 500, co-operation rate was 100% and our confidence interval was 97.5% with 5% margin of error. For quantitative data, mean and standard deviation were calculated. Qualitative results were calculated in percentages and presented in tabular forms.

ELIGIBILITY:
Inclusion Criteria:

* female sex, age ≥ 20 years, patients with availability of complete clinical details, biopsy proven breast cancer, no previous history of breast cancer treatment from other centers, males, all regional ethnicities(residents of Karachi, Sindh) and all stages of breast cancer

Exclusion Criteria:

* previously treated breast cancer patients, female ≤19 years, male/transgender, females coming for treatment for other provinces/foreigners.

Ages: 20 Years to 85 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Females were included in our study because more than 99% of our patients presenting with breast cancer were females, so we carried out our study on females only due to high prevalence rates
Study Population: 500 female patients were included in the study after taking informed written consent. All patients presented to single unit of a public sector hospital in Karachi, over the period of 10 years from 2010 till 2020.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Age | 10 years
  Age range assessed as compare to other studies and included range from 20 years till 85 years, because majority of cases fall in this category
Ethnicity | 10 years
  different ethnic groups residing in Karachi were assessed, based on city population data on different ethnicities living in the city
Stage of tumor at presentation | 10 years
  Staging of the tumor done according to NCCN guidelines
Breast cancer subtype | 10 years
  breast cancer subtype identified according to classification data available on subtypes, based on histopathology
Family History | 10 Years
  family history data acquired by asking direct questions through the patients. One or more positive relatives with breast cancer in the family were labelled as family history positive patients
Menopausal status | 10 year
  menopausal status was asked by patients if they not have had their last period since last 12 months. 12 months period criteria was set

SECONDARY OUTCOMES:
Risk factors, marital status, parity, symptoms, lump size and site at presentation | 10 years
  secondary outcomes were studied to look for relation of breast cancer with marital status, parity/number of children, symptoms, lump size and site on presentation

CONTACTS AND LOCATIONS:
Locations (1):
- Bahria University Medical and Dental College Karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: 1 year
Access Criteria: Everyone can access

REFERENCES:
- [Derived] Sultan N, Memon SA, Mooghal M, Wali S, Khan W, Tahseen H, Khan M, Monis D. Ethnic predisposition, risk factors and breast cancer presentation; a 10-year data. Single centered prospective cohort study from Karachi. Ann Med Surg (Lond). 2022 Sep 9;82:104612. doi: 10.1016/j.amsu.2022.104612. eCollection 2022 Oct. PMID 36268285